CLINICAL TRIAL: NCT01732692
Title: Multicenter Endoscopist-blinded Randomized Parallel-group Comparative Study to Assess Efficacy, Safety and Tolerance of Morning-only Dosing Compared to Control Split-dosing With Nocturnal Pause in MOVIPREP® Bowel Preparation Prior to Colonoscopy
Brief Title: Evaluation of the Efficacy, Safety and Tolerance of Experimental Morning-only MOVIPREP® Bowel Preparation in Comparison With Split-dose With Nocturnal Pause MOVIPREP® Bowel Preparation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Norgine BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MV-9999-301-RU; U1111-1135-2011 (Registry Identifier: WHO)
Record Dates: First submitted 2012-10-19; First posted 2012-11-26 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-04

CONDITIONS: Bowel Preparation Prior to Endoscopic, Radiological and Other Examinations as Well as to Surgical Procedures Which Require Empty Bowel.
Keywords: Bowel preparation, MOVIPREP®
MeSH Terms: interventions — MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MOVIPREP (Morning-only dose) (Experimental): MOVIPREP 250 ml solution every 15 minutes for up to one hour (4 doses in 1 hour=1 litre of solution), twice within same morning of colonoscopy.
  Interventions: Drug: MOVIPREP
- MOVIPREP (Split-dose) (Other): MOVIPREP 250 ml solution every 15 minutes for up to one hour (4 doses in 1 hour=1 litre of solution), once the evening before colonoscopy and once the morning of colonoscopy.
  Interventions: Drug: MOVIPREP

INTERVENTIONS:
Drug: MOVIPREP — MOVIPREP solution

SUMMARY:
To compare colon cleansing quality induced by the 2 different modes of MOVIPREP® intake in 5 colon segments prior to colonoscopy.

DETAILED DESCRIPTION:
All participants enrolled to the study will be allocated to one of two arms. Patients of the experimental morning-only regimen arm will prepare and take MOVIPREP® solution in the full dose - 2 litres of MOVIPREP® preparation in the early morning on the day of the colonoscopy clinical procedure. Participants in the standard split-dose regimen arm will prepare and take MOVIPREP® solution in split doses - ½ of dose (1 litre) the evening before + ½ of dose (1 litre) of MOVIPREP® preparation in the morning of the day of the colonoscopy.

The study consists of three visits. Participation in the study lasts no more than 11 days; 3 days as minimum.

There is no follow-up period planned except in case of any adverse events (AEs) when the follow-up period will last until the participant has recovered or until all AE-related queries for the participant have been resolved.

ELIGIBILITY:
Inclusion Criteria:

* male or female ≥18 years and ≤ 85 years
* colonoscopy procedure indicated
* willing to stay in the outpatient clinical site for colonoscopy and questionnaire completion
* willing and able to undergo study-related procedures
* informed consent signed by a patient for participation in the study
* negative pregnancy test in women with childbearing potential and consent for double barrier method birth control for subjects, men and women, during the study

Exclusion Criteria:

* ileus
* suspected colonic tumor with manifestations of intestinal obstruction
* delayed gastric emptying (gastroparesis), weak vomiting reflex, tendency to aspiration and regurgitation
* toxic megacolon which is a result of severe inflammatory conditions of the colon including Crohn's disease and ulcerative colitis
* suspected intestinal perforation or risk of gastrointestinal perforation
* signs of severe intestinal bleeding
* acute inflammatory anal or perianal pathology
* severe concomitant diseases of internal organs
* psychiatric diseases in aggravation stage
* hypersensitivity to polyethylene glycol and/or any component of MOVIPREP® preparation
* phenylketonuria or diagnosed glucose-6-phosphate dehydrogenate deficiency
* unconsciousness
* dehydration
* severe inflammatory diseases
* acute abdominal pain of unknown etiology
* pregnancy and lactation period
* participation in any other clinical study (including studies of experimental devices) in 30 days prior participation in the present trial
* patients who test positive for human immunodeficiency virus (HIV)/autoimmune disease (AID), Wasserman reaction (RW) or hepatitis B virus (HBC)
* any condition or circumstance that, in the opinion of the Investigator, would compromise the safety of the participant or the quality of study data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (3):
- Alma-Ata, Kazakhstan
- Russia (2):
  - Moscow
  - Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the Russian Federation and the Republic of Kazakhstan from 22 November 2012 to 5 April 2013.
Pre-assignment Details: Participants indicated for a colonoscopy were enrolled equally in 1 of 2 treatment groups, morning-only on the day of the clinical procedure or split-dosing in 2 stages with a nocturnal pause.
Period: Overall Study
Arm/Group | MOVIPREP (Morning-only Dose) | MOVIPREP (Split-dose)
Started | 70 | 70
Completed | 70 | 69
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MOVIPREP (Morning-only Dose) | MOVIPREP (Split-dose) | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (17.41) | 49.1 (16.26) | 49.8 (16.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 55 | 93
  Male | 32 | 15 | 47
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 4 | 10
  White | 64 | 66 | 130
Height [Mean (Standard Deviation); unit: cm] | 171.1 (9.36) | 165.1 (7.83) | 168.1 (9.07)
Weight [Mean (Standard Deviation); unit: kg] | 73.5 (16.92) | 68.3 (13.86) | 71.1 (15.75)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.1 (5.30) | 25.1 (5.10) | 25.1 (5.25)
Region of Enrollment [Number; unit: participants]
  Russia | 57 | 63 | 120
  Kazakhstan | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Colon Cleansing
Description: Bowel cleansing was assessed by a blinded endoscopist through visual evaluation of 5 colon segments and scored using the Harefield Cleansing Scale (HCS): A = success, all segments clean/scored 4 or 3; B = success, ≥1 segment with liquid/semi-solid amounts of stool, fully removable, ≥1 segment scored 2; C = failure, ≥1 segment with semi-solid or solid amounts of stool, at least 1 segment scored 1; and D = failure, ≥ 1 segment with irremovable, heavy, hard stools, ≥ 1 segment scored 0. Segmental evaluation of colon cleansing scores is as follows: 4: Colon empty and clean, no remaining stool or liquid. 3: Presence of clear liquid in the gut which can be removed by suction. 2: Brown liquid or semisolid remaining amounts of stool, fully removable. 1: Semisolid amounts of stool, only partially removable, difficult to make colonoscopy; 0: Irremovable, heavy, hard stools, colonoscopy impossible. Success of cleansing was defined as Grades of bowel cleansing А and В.
Time Frame: 1 day (the day of colonoscopy)
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | MOVIPREP (Morning-only Dose) | MOVIPREP (Split-dose)
Number analyzed (Participants) | 70 | 70
percentage of participants | 94.29 | 91.43
Statistical Analysis 1: Comparison: MOVIPREP (Morning-only Dose) vs MOVIPREP (Split-dose); Test type: Non-Inferiority or Equivalence — The primary endpoint was analyzed by a non-inferiority test using the exact Farrington-Manning method. Non-inferiority of the two treatments was to be concluded if the lower end of the confidence interval of the difference the experimental treatment group (morning-only dose) - control treatment group (split dose) was above a non-inferiority margin of -0.15%; p < 0.001, Exact Farrington - Manning; Treatment Difference = 0.0286, 95% CI 1-sided [lower limit -0.097] — Treatment Difference is the difference in proportion of participants with successful colon cleansing between treatments -experimental vs. control

2. Secondary Outcome: Patient Satisfaction of Colonoscopy Preparation (VAS)
Description: Patient satisfaction was measured on a 100 mm visual analog scale (VAS) where 0 (left end of the line) is marked as "totally unacceptable" (lowest patient satisfaction of colonoscopy preparation) and 100 is "fully acceptable" (highest patient satisfaction with the procedure). Satisfaction was scored based on a mark placed on the line by the participant.
Time Frame: 1 day (the day of colonoscopy)
Population: Intent-to-treat population with available VAS data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOVIPREP (Morning-only Dose) | MOVIPREP (Split-dose)
Number analyzed (Participants) | 70 | 69
units on a scale | 81.2 (20.97) | 79.6 (23.18)

3. Secondary Outcome: Total Compliance Score
Description: Compliance score = 100 * (total amount MOVIPREP® intake) / (planned MOVIPREP intake).
  Total compliance score of MOVIPREP is the average score of the compliance for the first and second litre.
Time Frame: 1 day (the day of colonoscopy)
Population: Intent-to-treat with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOVIPREP (Morning-only Dose) | MOVIPREP (Split-dose)
Number analyzed (Participants) | 70 | 69
units on a scale | 98.1 (6.10) | 99.5 (2.66)

4. Secondary Outcome: Patient Compliance - Amount of Additional Clear Liquid Consumed
Description: To prevent any potential dehydration risk participants were recommended the intake of at least 500 ml of additional clear liquid (juices without pulp, tea, water) per liter of the Moviprep solution. The amount of additional clear liquid taken is reported for each liter of Moviprep taken.
Time Frame: 1 day (the day of colonoscopy)
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | MOVIPREP (Morning-only Dose) | MOVIPREP (Split-dose)
Number analyzed (Participants) | 70 | 69
ml
  After first liter of study drug | 545.43 (128.6) | 640.29 (243.4)
  After second liter of study drug | 539.71 (116.5) | 585.65 (145.2)

5. Secondary Outcome: Percentage of Patients Who Experienced Adverse Events (AEs)
Description: An AE was a worsening in severity or frequency of a concomitant illness or any new illness diagnosed during the clinical trial period. A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability / incapacity; is a congenital anomaly / birth defect; is medically important. Severity is a clinical observation and describes the intensity of the event: Mild: Transient symptoms, no interference with daily activities; Moderate: Marked symptoms, moderate interference with daily activities; Severe: Considerable interference with daily activities. Relatedness to study drug was assessed by the Investigator.
Time Frame: From first dose of study drug until the end of colonoscopy procedure, maximum of 24 hours.
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | MOVIPREP (Morning-only Dose) | MOVIPREP (Split-dose)
Number analyzed (Participants) | 70 | 70
percentage of participants
  Any adverse event (AE) | 58.6 | 61.4
  Mild adverse event | 52.9 | 54.3
  Moderate adverse event | 5.7 | 7.1
  Severe adverse event | 0.0 | 0.0
  Serious adverse event | 0.0 | 0.0
  AE leading to study discontinuation | 0.0 | 1.4
  Treatment-related adverse event | 57.1 | 58.6

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until the end of the colonoscopy, maximum of 24 hours.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | MOVIPREP (Morning-only Dose) | MOVIPREP (Split-dose)
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 41/70 | 43/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOVIPREP (Morning-only Dose) (N=70) | MOVIPREP (Split-dose) (N=70)
Abdominal discomfort (Gastrointestinal disorders) | 13 | 26
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Abdominal tenderness (Gastrointestinal disorders) | 1 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 30 | 22
Vomiting (Gastrointestinal disorders) | 5 | 7
Product taste abnormal (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood calcium decreased (Investigations) | 0 | 1
Blood calcium increased (Investigations) | 1 | 0
Blood chloride increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 1
Blood glucose increased (Investigations) | 3 | 0
Blood iron decreased (Investigations) | 1 | 5
Blood iron increased (Investigations) | 2 | 1
Body temperature increased (Investigations) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.